CLINICAL TRIAL: NCT04958525
Title: A Controlled Observational Study on Minimally Invasive Treatment of Hypertensive Basal Ganglia Hemorrhage by Transfrontal Keyhole Neuroendoscopy
Brief Title: Minimally Invasive Treatment of Hypertensive Basal Ganglia Hemorrhage by Transfrontal Keyhole Neuroendoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020543
Record Dates: First submitted 2021-06-28; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Basal Ganglia Hemorrhage
Keywords: Hypertensive basal ganglia hemorrhage; Transfrontal keyhole neuroendoscopic technique; Ultrasonic positioning
MeSH Terms: conditions — Basal Ganglia Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic Surgery Group: After a full evaluation of the patient's condition, the informed consent was signed to perform keyhole neuroendoscopic ultrasound-guided hematoma removal for the patient.
  Interventions: Procedure: Keyhole neuroendoscopic transfrontal ultrasound-guided hematoma removal
- Microsurgery group: After a full evaluation of the patient's condition, the informed consent was signed to perform small bone window craniotomy for hematoma removal under microscope for the patient.
  Interventions: Procedure: Small bone window craniotomy for hematoma removal under microscope

INTERVENTIONS:
Procedure: Keyhole neuroendoscopic transfrontal ultrasound-guided hematoma removal — Keyhole neuroendoscopic transfrontal ultrasound-guided hematoma removal in basal ganglia region:According to the brain CT scan and reconstruct the operation plan, choose a side by 2 cm before the coronal suture line 4 cm and 3 cm center longitudinal incision formation of 2 cm bone drilling the hole, ultrasonic measurement and the size of hematoma puncture depth, and guide the puncture direction, the transparent channel under endoscopic direct placement hematoma backend, after entering the hematoma cavity, under the neural endoscopic removal of hematoma,Wash the hematoma cavity with warm salt water.Bipolar electrocoagulation hemostasis for active bleeding.An indwelling drainage tube was placed in the hematoma cavity, and ultrasonography determined that the hematoma was cleared satisfily without active bleeding.
  Groups: Endoscopic Surgery Group
Procedure: Small bone window craniotomy for hematoma removal under microscope — Small bone window craniotomy for hematoma removal under microscope:Small bone window craniotomy in frontotemporal region, no blood vessels and non-functional areas of the hematoma nearest to the cortex was cut open, the hematoma was removed under the microscope and the cavity of the hematoma was washed with warm saline, and bipolar electrocoagulation hemostasis was performed for active bleeding.An indwelling drainage tube was placed in the hematoma cavity and the operation was completed without active bleeding.
  Groups: Microsurgery group

SUMMARY:
To compare the prognosis of patients with hypertensive intracerebral hemorrhage treated by two different surgical methods, and to clarify the therapeutic effect of minimally invasive surgery, so as to find a better surgical method that can reduce surgical trauma and mortality and improve the prognosis of patients

DETAILED DESCRIPTION:
In this study, a cohort observation method was adopted to observe a total of 52 patients who underwent two surgical procedures, namely, removal of hematoma in basal ganglo-region by keyhole neuroendoscopy under frontal ultrasound guidance and removal of hematoma by craniotomy microsurgery. They were divided into the endoscopic surgery group and the microsurgery group. In the endoscopic surgery group, 26 patients underwent removal of hematoma in basal ganglo-region by keyhole neuroendoscopy under frontal ultrasound guidance.In the microsurgery group, 26 cases were treated with craniotomy microsurgery for hematoma removal. The clearance rate of surgical hematoma, surgical safety, GCS score, GOS score, nerve fiber injury and postoperative complications were observed in the two groups 1 week, 1 month and 3 months after surgery.To observe and analyze whether endoscopic surgery group has advantages in improving hematoma clearance rate and efficacy

ELIGIBILITY:
Inclusion Criteria:

* CT scan was used to diagnose cerebral hemorrhage in basal ganglia region. The amount of bleeding was 30-50ml, and no cerebral hernia was formed.
* Age between 30 and 70
* The onset is longer than 24 hours and less than 72 hours.
* Informed consent of the patient and/or their relative.

Exclusion Criteria:

* Brain injury, hemorrhage caused by intracranial aneurysm or cerebral arteriovenous malformation.
* Coagulation dysfunction
* Insufficiency of vital organs of heart, liver, kidney or lung
* Previous history of stroke with functional loss
* Intracranial or systemic infection
* Poor blood pressure control

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients from Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Hemorrhage clearance evaluation | 3 months after surgery was done
  Preoperative and postoperative hematoma volume and hematoma clearance rate were evaluated by cerebral fibrous tract imaging
Prognosis of Minimally Invasive Treatment of Hypertensive Basal Ganglia Hemorrhage | 3 months after surgery was done
  Glasgow coma score (GCS) score, GOS score, 1 month postoperative mortality, and 7 days postoperative complications were evaluated: gastrointestinal stress ulcer bleeding, intracranial infection.Mortality and Glasgow and GOS scores at 30 days and 3 months after surgery were evaluated by telephone interviews or inpatient records.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Bin, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No